CLINICAL TRIAL: NCT06663891
Title: Identification of Trait Markers Differentiating Late-onset Depression from Early-onset Depression in Chronic Anergic Depression in the Elderly
Brief Title: Chronic Anergic Depression IDentification - Magnetic Resonance Imaging Exploration in the Elderly of Traits Related to Onset
Acronym: CAnD'ID-METRO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9203; 2024-A02236-41 (Other: ANSM)
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Late Life Depression
Keywords: Late life depression neuroimaging,; connectivity,; apathy,; dopaminergic system
MeSH Terms: conditions — Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Onset Depression (EOD) (Other): Elderly depressed patients (≥ 60 years and < 90 years) suffering from active or remitted anergic depression and who have at least one history of a depressive episode strictly before the age of 60 years
  Interventions: Other: Functional MRI with EEG per MRI
- Late Onset Depression (LOD) (Other): Elderly depressed patients (≥ 60 years and < 90 years) suffering from active or remitted anergic depression and who do not have a history of a depressive episode strictly before the age of 60 years.
  Interventions: Other: Functional MRI with EEG per MRI

INTERVENTIONS:
Other: Functional MRI with EEG per MRI — 2 MRI examinations will be carried out on a Siemens Vida® MRI ( Siemens®, Erlangen, Germany) 3 Tesla. During this study, no MRI examination requires the injection of a contrast agent.
  Different sequences, according to several acquisition modalities, will be performed during each MRI. The structural sequences (T1 and T2, MPRAGE) will highlight any lesions in the form of atrophies and/or vascular lesions in the participants, also subject to inter-individual differences. The examination will also involve a quantitative multiparametric acquisition with 8 modalities (R1, R2, Radial and Axial Diffusion in Diffusion Tensor, dispersion, orientation and density index of neurites by NODDI, the Macromolecular Proton Fraction, measurement of magnetic susceptibility and R2*) to characterize tissue properties. Functional imaging (in resting state, during film viewing and performance of cognitive tasks in ASL, BOLD and multiband) will allow analysis of the primary endpoint - functional connectivity,

SUMMARY:
Depression in the elderly, or "late life depression" (LLD), is often considered to be homogeneous, legitimizing standardized treatment. Yet the literature suggests that there are different forms of LLD, with different pathophysiology, course and treatment.

Our experience has led us to identify an "anergic" form, marked by adynamia and anhedonia (anergic depression, AnD). Highly represented among LLDs, it readily resists the usual antidepressants, so that its course is often chronic. Thanks to the "Chronic Anergic Depression Open Trial", the investigators were able to show that AnD responds to dopaminergic (DA) molecules. Therefore the invastigators hypothesized a pathophysiology linked to dysfunction of the mesolimbic DA system.

However, not all patients would present the same form: two subgroups could be isolated, each contributing equally. The first corresponds to patients for whom the episode is a recurrence, the so-called "early onset depression" (EOD). The first episode occurs at 34 ±16 years of age and is frequently associated with a personality disorder (73%). The index episode usually lasts 6 ±3 years and is typically associated with anxiety (96%).

The second group corresponds to the onset of primary depression after the age of 60, known as "late onset depression" (LOD). The index episode occurs at around 71 ±6 years of age, in people with no premorbid personality disorders. The episode is shorter (3 ±1 years) and anxiety is frequent (75%) but less marked. These patients showed a high propensity for a course compatible with synucleinopathies, but often less rapid than that of the classic forms of these diseases.

The investigators hypothesize that within AnD, EOD and LOD present different pathophysiologies, and that this difference is observable on functional magnetic resonance imaging (MRI): LOD patients should present a greater reduction in functional connectivity in the mesolimbic system. The investigators make the subsidiary hypothesis that LODs also show a structural alteration observable with other types of MRI measurements, i.e. multiparametric imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 60 (inclusive) to 90 years (exclusive)
* Patient presenting with active or remitted anergic depression according to the operational criteria of the "Chronic Anergic Depression Open Trial" (1) confirmed by two psychiatrists involved in the study:

  * Early Onset Depression (EOD) group: with at least one history of depression before age 60
  * Late Onset Depression (LOD) group: no history of depression before age 60
* Patient able to understand the objectives/risks of the research and give informed consent
* Patient affiliated to a health insurance social protection scheme, beneficiary or dependent

Exclusion Criteria:

* Contraindication to an MRI scan (including claustrophobia)*
* Psychiatric or organic comorbidity that may interfere with the interpretation of results (e.g. neurovascular disease, psychotic disorder, proven neurodegenerative disease)
* Concomitant treatment that may interfere with the interpretation of results (e.g. interferons, corticosteroids)
* Patient in exclusion period (from a previous or current study)
* Current protective measure (curatorship, guardianship)
* Patient under legal protection * presence of non-removable ferromagnetic foreign body, prosthesis, pacemaker, defibrillator, neurostimulation device, medications delivered by an implanted pump, vascular clip or stent, heart valve or ventricular shunt, implanted device incompatible with 3 Tesla MRI exam, claustrophobia, epilepsy

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
VTA - mesolimbic system functional connectivity | Day 1
  Functional connectivity, observed at the subpopulation level, between the ventral tegmental area (VTA) and regions of the mesolimbic system (i.e.: ventral striatum and pallidum, amygdala, and subgenual anterior cingulate [with separate analysis of Brodmann area 25] and ventromedial prefrontal cortex), obtained by ROI to ROI analysis.

SECONDARY OUTCOMES:
Perfusion of the mesolimbic system | Day 1
  Mean cerebral perfusion rates measured by arterial spin labeling (ASL) in regions of interest (i.e.: ventral tegmental area, ventral striatum and pallidum, amygdala, and subgenual anterior cingulate [with separate analysis of Brodmann area 25] and ventromedial prefrontal cortex).
Perfusion of the mesolimbic system | Day 13
  Mean cerebral perfusion rates measured by arterial spin labeling (ASL) in regions of interest (i.e.: ventral tegmental area, ventral striatum and pallidum, amygdala, and subgenual anterior cingulate [with separate analysis of Brodmann area 25] and ventromedial prefrontal cortex).

OTHER OUTCOMES:
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  R1
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  R1
Θ / β powers ratio | Day 1
  Frequency and maximum intensity of fluctuations in the ratio between the powers in θ and β bands. This analysis aims to allow the localization of the regions associated with fluctuations in vigilance during acquisition. This localization will be allowed by a methodology and analysis parameters already published by our team. The MRI localization maps obtained at the subpopulation level will be compared.
Θ / β powers ratio | Day 13
  Frequency and maximum intensity of fluctuations in the ratio between the powers in θ and β bands. This analysis aims to allow the localization of the regions associated with fluctuations in vigilance during acquisition. This localization will be allowed by a methodology and analysis parameters already published by our team. The MRI localization maps obtained at the subpopulation level will be compared.
Mesolimbic system - whole brain functional connectivity | Day 1
  Functional connectivity, observed at the subpopulation level, between regions of the mesolimbic system (as defined according to the primary outcome measure) and the rest of the brain, obtained by seed-to-voxel analysis.
  The seeds will be the regions of the mesolimbic system (i.e.: the ventral striatum and pallidum, the amygdala, the subgenual anterior cingulate cortex [with separate analysis of Brodmann area 25] and ventromedial prefrontal cortex and the substantia nigra). The analysis area will be the entire brain .
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  Radial and Axial Diffusion in Diffusion Tensor
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  R2
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  R2
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  Radial and Axial Diffusion in Diffusion Tensor
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  Dispersion index
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  Dispersion index
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  Orientation and density of neurites by NODDI
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  Orientation and density of neurites by NODDI
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  Macromolecular Proton Fraction
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  Macromolecular Proton Fraction
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 1
  Measurement of magnetic susceptibility and R2
Quantitative parameters measured in multiparametric MRI in the ventral tegmental area | Day 13
  Measurement of magnetic susceptibility and R2

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic DORMEGNY-JEANJEAN Doctor, Principal Investigator — Department of Physiology and Funtional Explorations at Strasbourg University Hospitals

IPD SHARING:
Plan to Share IPD: No